CLINICAL TRIAL: NCT05983757
Title: A Phase III, Randomized, Multicenter, Investigational, Open Label Clinical Trial That Will Examine Whether Treatment With Endovascular Thrombectomy is Superior to Standard Medical Therapy Alone in Patients Who Suffer a Distal Medium Vessel Occlusion Ischemic Strokes.
Brief Title: Combined Thrombectomy for Distal MediUm Vessel Occlusion StroKe
Acronym: DUSK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Raul Nogueira (Other)
Collaborators: Stryker Neurovascular (Industry); Brainstorme Imaging Core Lab Inc (Unknown)
Responsible Party: Sponsor-Investigator, Raul Nogueira, Director, UPMC Stroke Institute, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY23030032
Record Dates: First submitted 2023-07-20; First posted 2023-08-09 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Ischemic
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Intervention Model Description: The randomization employs a 1:1 ratio of endovascular thrombectomy (EVT) with the use of Trevo NXT ProVue Retrievers, AXS Vecta 46 Intermediate Catheter and AXS Catalyst 5 Distal Access Catheter, versus standard medical management (SMM) in patients who suffer a distal medium vessel occlusion (DMVO) stroke within 12 hours from time last seen well (TLSW) and have evidence of salvageable brain tissue on perfusion imaging. Randomization will be done under a minimization process using age (≤67 vs. >67 years), baseline NIHSS (≤12 vs. >12), use of IV thrombolysis (none vs. within 120 minutes from randomization vs. > 120 minutes from randomization), site of occlusion (M2 vs. M3 vs. ACA vs. PCA), baseline infarct volume (≤15mL vs. >15-30mL vs. >30-50mL), perfusion mismatch volume (≤15mL vs. >15-30mL vs. >30-50mL), therapeutic window (0-4.5 vs. 4.5-8 or >9-12 hours after TLKW), and participating site.
Who Masked: Outcomes Assessor
Masking Description: One investigator or designee will remain blinded at each site to perform primary outcome assessment at Day 30 and Day 90.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care Treatment (Active Comparator): Standard medical management in patients who suffer a distal medium vessel occlusion
  Interventions: Other: Standard medical management
- Endovascular Thrombectomy (Experimental): Endovascular thrombectomy in patients who suffer a distal medium vessel occlusion.
  Interventions: Device: Experimental: endovascular thrombectomy in patients who suffer a distal medium vessel occlusion

INTERVENTIONS:
Device: Experimental: endovascular thrombectomy in patients who suffer a distal medium vessel occlusion — The AXS Catalyst Distal Access Catheter is indicated for use in facilitating the insertion and guidance of appropriately sized interventional devices into a selected blood vessel in the peripheral and neurovascular systems, and is also indicated for use as a conduit for retrieval devices.
  The AXS Vecta Intermediate Catheter, as part of the AXS Vecta Aspiration System, is indicated in the revascularization of patients with acute ischemic stroke. Patients who are ineligible for intravenous tissue plasminogen activator (IV t-PA) or who failed IV t-PA therapy are candidates for treatment.
  The Trevo® Retriever is indicated for use to restore blood flow in the neurovasculature by removing thrombus for the treatment of acute ischemic stroke to reduce disability in patients with a persistent, proximal anterior circulation, large vessel occlusion, and smaller core infarcts who have first received intravenous tissue plasminogen activator (IV t-PA).
  Other Names: AXS Vecta 46; AXS CAT 5; NXT ProVue Retriever
  Arms: Endovascular Thrombectomy
Other: Standard medical management — All subjects should receive the best standard medical therapy based on current AHA guidelines. Subjects randomized to standard medical management (SMM) will receive standard medical therapy only based on the guidelines. All subjects are expected to be admitted to hospital as part of routine best guideline-based care and treated on a stroke unit or neurointensive care unit or equivalent.
  Other Names: Active Comparator
  Arms: Standard of Care Treatment

SUMMARY:
A phase III, randomized, multi-center, investigational, open label clinical trial that will examine whether treatment with endovascular thrombectomy is superior to standard medical therapy alone in patients who suffer a Distal Medium Vessel Occlusion Ischemic Stroke within 12 hours from time last seen well

DETAILED DESCRIPTION:
DUSK is a Phase-3, prospective, multicenter, investigational, randomized, controlled, open-label study with blinded endpoint evaluation (PROBE design) and an adaptive design with population enrichment. The randomization employs a 1:1 ratio of endovascular thrombectomy (EVT) versus standard medical management (SMM) in patients who suffer a distal medium vessel occlusion (DMVO) stroke within 12 hours from time last seen well (TLSW) and have evidence of salvageable brain tissue on perfusion imaging. Randomization will be done under a minimization process using age (≤67 vs. >67 years), baseline NIHSS (≤12 vs. >12), use of IV thrombolysis (none vs. within 120 minutes from randomization vs. > 120 minutes from randomization), site of occlusion (M2 vs. M3 vs. ACA vs. PCA), baseline infarct volume (≤15mL vs. >15-30mL vs. >30-50mL), perfusion mismatch volume (≤15mL vs. >15-30mL vs. >30-50mL), therapeutic window (0-4.5 vs. 4.5-8 or >9-12 hours after TLKW), and participating site. The candidate enriched populations that the trial considers are based on use of intravenous thrombolysis (none vs. within 120 minutes from randomization vs. > 120 minutes from randomization), TLKW to randomization (0-6 vs. 6-12 hours) and mismatch volumes as measured using absolute mismatch (defined as Tmax>6 sec - DWI lesion on MRI or Tmax>6 sec -rCBF<30% lesion on CTP) (>40 cc vs. >30cc vs. >20cc vs. >10cc). The primary endpoint will be a categorical shift across all levels on the modified Rankin Scale (mRS) at 90-days post-randomization. The hypothesis is that EVT will lead to an improved clinical outcome at 90 days. Interim analysis will be performed after the primary endpoint is available for a total of 386 randomized patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years (no upper age limit)
2. Acute ischemic stroke where patient is ineligible for or has failed* IV thrombolytic treatment and is ineligible for endovascular treatment under best guideline-based care due to absence of proximal arterial occlusion (e.g. intracranial ICA, MCA-M1 and co-dominant or dominant M2** segments, and vertebrobasilar arteries).***

   * IV thrombolytic treatment failure is defined by persistent disabling neurological deficits beyond 60 minutes of completion of thrombolytic infusion in the presence of imaging findings consistent with DMVO.

   **Dominant M2 segment is defined is a division supplying >50% of the MCA territory vs co-dominant supplying 50% of the MCA territory vs non-dominant supplying <50% of the MCA territory.

   ***No procedures or tests required by the protocol will delay fastest possible delivery of thrombolytic therapy to potentially eligible subjects.
3. Evidence of a primary (e.g. not secondary to EVT of proximal vessel occlusion) distal medium vascular occlusion defined as occlusion of the non-dominant M2 segment or M3 segment of the MCA, the ACA (A1, A2, or A3 segments), or the PCA (P1, P2 or P3 segments) resulting in significant clinical deficits and expected to be treatable by endovascular thrombectomy. Regardless of vessel anatomic location, all vessel diameters should be within 1.5mm -2.5mm. (refer to the device labeling for recommended vessel diameters for each device model.)*
4. No significant pre-stroke functional disability (mRS ≤2)
5. Evidence of a disabling stroke defined as follows:

   1. Baseline National Institutes of Health Stroke Scale (NIHSS) score >5 at the time of randomization.
   2. NIHSS 3-5 with disabling deficit including significant aphasia, neglect, hemianopsia, or hemiparesis/ loss of hand or leg function as established by the treating team in context of the patient's life.
6. The presence of a Target Mismatch defined as:

   1. Ischemic Core < 50cc (defined on NCCT/CTP* or DWI-MRI)

      *Visual or automatedly detected hypodensity on NCCT should be used to exclude or include patients if the investigator believes that their assessment is more reliable than the CTP volume in any particular case.
   2. Mismatch Volume (TMax >6sec lesion - Core volume lesion) >10cc
   3. Mismatch Ratio >1.4
7. Patient treatable within 12 hours of symptom onset. Symptoms onset is defined as the point in time the patient was last seen well (at baseline). Treatment start is defined as the time of arterial puncture.
8. Informed consent obtained from patient or acceptable patient surrogate

Exclusion Criteria:

1. Any sign of intracranial hemorrhage on baseline CT/MR (SDH/SAH/ICH).
2. Rapidly improving symptoms, particularly if in the judgment of the managing clinician that the improvement is likely to result in the patient having no residual disabling deficits and an NIHSS score of <5 at randomization.
3. Significant ischemic changes in a territory other than the occluded site that in the opinion of the investigator could reduce the benefit of endovascular treatment.
4. Contra indication to imaging with MR or CT with contrast agents.
5. Infarct core >1/3 occluded territory (MCA, ACA, or PCA) qualitatively or >50 mL quantitatively (determined by NCCT, CTP or DWI).
6. Any terminal illness such that patient would not be expected to survive more than 1 year.
7. Recent past history or clinical presentation of ICH, subarachnoid hemorrhage (SAH), arterio-venous (AV) malformation, aneurysm, or cerebral neoplasm other than meningioma.
8. Any imaging findings suggestive of futile recanalization in the judgment of the local investigator.
9. Premorbid disability (mRS ≥3).
10. Inability to initiate endovascular treatment within 12 hours of last seen well.
11. Seizures at stroke onset if it precludes obtaining an accurate baseline NIHSS.
12. Baseline blood glucose of <50 mg/dL (2.78 mmol) or >400 mg/dL (22.20 mmol).
13. Known history of hereditary or acquired hemorrhagic diathesis and/or platelet count <100,000/uL.
14. Known renal failure as defined as serum creatinine levels > 3.0 mg/dL.
15. Presumed septic embolus or suspicion of bacterial endocarditis.
16. Any other condition that, in the opinion of the investigator, precludes an endovascular procedure or poses a significant hazard to the subject if an endovascular procedure was performed.
17. History of drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
18. Subjects with occlusions in multiple vascular territories (e.g., bilateral or multi-territorial anterior circulation, or anterior/posterior circulation)
19. Subject participating in a study involving an investigational drug or device that would impact this study
20. Known pregnancy
21. Prisoner or incarceration
22. Known acute symptomatic COVID-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Shift in distribution of all levels of the 90-day modified Rankin Scale with levels 5-6 combined (mRS; 0, 1, 2, 3, 4, 5-6) as assessed by structured assessment | 90-day follow-up
  Modified Rankin Scale measurement (mRS): 0=no symptoms, 1= no significant disablity despite symptoms, able to carry out all usual duties. 2= slight disability, unable to carry out all previous activities, but able to look after own affairs without assistance. 3=moderate disability, requiring some help, able to walk without assistance. 4=moderatly severe disability, unable to walk and attend to bodily needs without assistance. 5=severe disability, bedridden, incontinent and requiring total nursing care. 6=dead

SECONDARY OUTCOMES:
Shift in distribution of the 90-day mRS (0;1;2;3;4;5;6) as assessed by structured assessment | 90-day follow-up
  Modified Rankin Scale measurement (mRS)0=no symptoms, 1= no significant disablity despite symptoms, able to carry out all usual duties. 2= slight disability, unable to carry out all previous activities, but able to look after own affairs without assistance. 3=moderate disability, requiring some help, able to walk without assistance. 4=moderatly severe disability, unable to walk and attend to bodily needs without assistance. 5=severe disability, bedridden, incontinent and requiring total nursing care. 6=dead
Rates of Independent Outcome defined as mRS ≤2 and/ or equal to Baseline mRS at 90 days | 90-day follow-up
  Independant outcome: 0=no symptoms, 1= no significant disablity despite symptoms, able to carry out all usual duties. 2= slight disability, unable to carry out all previous activities, but able to look after own affairs without assistance. 3=moderate disability, requiring some help, able to walk without assistance. 4=moderatly severe disability, unable to walk and attend to bodily needs without assistance. 5=severe disability, bedridden, incontinent and requiring total nursing care. 6=dead
Rates of Excellent Outcome defined as mRS ≤1 and/ or equal to Baseline mRS at 90 days | 90-day follow-up
  Excellent outcome: 0=no symptoms, 1= no significant disablity despite symptoms, able to carry out all usual duties. 2= slight disability, unable to carry out all previous activities, but able to look after own affairs without assistance. 3=moderate disability, requiring some help, able to walk without assistance. 4=moderatly severe disability, unable to walk and attend to bodily needs without assistance. 5=severe disability, bedridden, incontinent and requiring total nursing care. 6=dead.
Rates of Good Functional Outcomes adjusted for the baseline mRS and stroke severity (NIHSS) according to the modified Rankin Scale scores at 90 days as following: | 90-day follow-up
  NIHSS and mRS scores MRS: 0=no symptoms, 1= no significant disablity despite symptoms, able to carry out all usual duties. 2= slight disability, unable to carry out all previous activities, but able to look after own affairs without assistance. 3=moderate disability, requiring some help, able to walk without assistance. 4=moderatly severe disability, unable to walk and attend to bodily needs without assistance. 5=severe disability, bedridden, incontinent and requiring total nursing care. 6=dead NIHSS: 0=no stroke symptoms, 1-4=minor stroke, 5-15 moderate stroke, 16-20 moderate to sever stroke, 21-42- severe stroke.
  * If NIHSS <10 and Baseline mRS 0 or 1: 90-day mRS ≤1
  * If NIHSS <10 and Baseline mRS 2: 90-day mRS ≤2
  * If NIHSS ≥10 and Baseline mRS 0 or 1: 90-day mRS ≤2
  * If NIHSS ≥10 and Baseline mRS 2: 90-day mRS ≤3
EVT arm only: Final reperfusion grades according to the extended Thrombolysis in Cerebral Infarction (eTICI) scale and the rates of First Pass Effect (eTICI ≥2c) and Modified First Pass Effect (eTICI ≥2b50) | 90-day follow-up
  Reprofusion grades :TICI scores:grade 0: no perfusion noted (0% reperfusion) grade 1: reduction in thrombus but without any resultant filling of distal arterial branches grade 2 grade 2a: reperfusion of 1-49% of the territory grade 2b50: reperfusion of 50-66% of the territory grade 2b67: reperfusion of 67-89% of the territory grade 2c: extensive reperfusion of 90-99% of the territory grade 3: complete or full reperfusion (100% reperfusion).
EVT arm only: Final reperfusion grades according to the rates of First Pass Effect (eTICI ≥2c) | 90-Day follow up
  Reprofusion grades :TICI scores:grade 0: no perfusion noted (0% reperfusion) grade 1: reduction in thrombus but without any resultant filling of distal arterial branches grade 2 grade 2a: reperfusion of 1-49% of the territory grade 2b50: reperfusion of 50-66% of the territory grade 2b67: reperfusion of 67-89% of the territory grade 2c: extensive reperfusion of 90-99% of the territory grade 3: complete or full reperfusion (100% reperfusion).
EVT arm only: Final reperfusion grades according to the Modified First Pass Effect (eTICI ≥2b50) | 90 day follow up
  Reprofusion grades :TICI scores:grade 0: no perfusion noted (0% reperfusion) grade 1: reduction in thrombus but without any resultant filling of distal arterial branches grade 2 grade 2a: reperfusion of 1-49% of the territory grade 2b50: reperfusion of 50-66% of the territory grade 2b67: reperfusion of 67-89% of the territory grade 2c: extensive reperfusion of 90-99% of the territory grade 3: complete or full reperfusion (100% reperfusion).
Mean score for disability on the utility-weighted modified Rankin scale (UW-mRS) at 90 days | 90-day follow-up
  utility weighted mRS 0=no symptoms, 1= no significant disablity despite symptoms, able to carry out all usual duties. 2= slight disability, unable to carry out all previous activities, but able to look after own affairs without assistance. 3=moderate disability, requiring some help, able to walk without assistance. 4=moderatly severe disability, unable to walk and attend to bodily needs without assistance. 5=severe disability, bedridden, incontinent and requiring total nursing care. 6=dead
Final infarct volume (FIV) (FIV - baseline infarct on CTP or DWI) evaluated on CT or MRI at 24 hours (-2/+12 hours) | 24 hours (-2hours /+12 hours)
  Infarct volume at 24 hours will be measured on CT or MRI.
Final infarct growth (FIV - baseline infarct on CTP or DWI) | 24 hours (-2 hours/+12 hours)
  Infarct volume at 24 hours will be measured on CT or MRI, growth of infarct from baseline to 24 hours will be captured.
Final infarct volume (FIV) and infarct growth (FIV - baseline infarct on CTP or DWI) evaluated on CT or MRI at 3-5 days (if available) | 3-5 days
  Infarct volume at 3-5 days will be measured on CT or MRI.
Final infarct growth (FIV - baseline infarct on CTP or DWI) evaluated on CT or MRI at 3-5 days (if available) | 3 to 5 days
  Infarct volume at 3-5 days will be measured on CT or MRI, growth of infarct will be compared to baseline.
Clinical improvement at 24 hours calculated as the difference between 24-hour and baseline NIHSS score | 24 hours
  NIHSS score at 24hours :NIHSS: 0=no stroke symptoms, 1-4=minor stroke, 5-15 moderate stroke, 16-20 moderate to sever stroke, 21-42- severe stroke.
Cost effectiveness analysis of endovascular thrombectomy vs standard medical therapy | 90-day follow-up
  Assessment of costs from the time of randomization to the 90 day follow up. This includes Costs of hospitalization, institutional living and outpatient care will be assessed and compared for each arm.
Brain tissue reperfusion evaluated by CT or MRI perfusion at 24 hours in both treatment groups (if available) | 24 hours
  CT or MRI results at 24 hours
Vessel patency evaluated by CTA or MRA perfusion at 24 hours in both treatment groups (if available) | 24 hours
  CTA or MRA perfusion results at 24 hours
Patient reported outcomes (EQ-5D) | 90-day follow-up
  Questionnaires assessed by blinded assessor at 90 days. EQ-5D measures mobility, self care, usual activities, pain and anxiety, overall heath is measured on a scale of 0 (worst health state) to 100 best health state.
Patient reported outcomes (PROMIS Global-10) | 90 day follow up
  Questionnaires assessed by blinded assessor at 90 days. Promise Global Health measures current health status on a scale of 1=poor, 2=fair, 3=good, 4=very good, 5=excellent. The scale is from 1-5 with 1 being the poorest health outcome and 5 the best.
Patient reported outcomes (PROMIS Fatigue) | 90 day follow up
  Questionnaires assessed by blinded assessor at 90 days. Promise Fatigue will measure degree of fatigue on a scale of 1=not at all, 2=a little bit, 3=somewhat, 4= quite a bit, 5=very much. The scale is from 1-5 with 1 being the least fatigued and 5 the greatest feeling of fatigue.
Patient reported outcomes ( IADL) | 90 day follow up
  Questionnaires assessed by blinded assessor at 90 days. IADL measures the ability to use a telephone, shop prepare food, do housekeeping, laundry, mode of transportation, medications and handle finances. The subject will answer the questions and answer as for how they are able to accomplish their ADLs.
Patient reported outcomes ( MoCa) | 90 day follow up
  Questionnaires assessed by blinded assessor at 90 days. MoCa measures the patient's ability to draw(visuospatial), name items, memory, attention, language, and abstraction. There are several questions that the subject will answer for each category.
All cause mortality | 90 day follow up
  All-cause mortality within 90 days
Mortality due to stroke | 90 day follow up
  Mortality within 90 days due to index stroke
Intracranial hemorrhage | 90 day follow up
  Symptomatic intracranial hemorrhage (SICH) defined as per the Heidelberg Classification: new intracranial hemorrhage detected by brain imaging associated with any of the item below:
  * ≥4 points total NIHSS at the time of diagnosis compared to immediately before worsening.
  * ≥2 point in one NIHSS category.
  * Absence of alternative explanation for deterioration. This will be the primary definition for SICH as per the recommendation of both the FDA and DSMB.
    * Symptomatic intracranial hemorrhage (SICH) defined as per the modified SITS-MOST definition.
Intracranial hemorrhage | 24 hours (-2 hours /+12 hours)
  The incidence of any intracranial hemorrhage measured at 24 (-2/+12) hours as graded by the central core-lab using the Heidelberg classification criteria.
Procedure-related vessel perforation. | 24 hours (-2 hours /+12 hours)
  Perforation of the artery related to the procedure.
Procedure-related vessel dissection | 24 hours (-2 hours/+12 hours)
  Dissection of an artery related to the procedure.
Embolization to a new territory during mechanical thrombectomy (MT) procedure | 24 hours (-2 hours/+12hours)
  New emboli to a different area of the brain during the MR procedure.
Significant extracranial hemorrhage (e.g., access site, retroperitoneal hematoma) requiring blood transfusion and/or surgical intervention. | 24 hours (-2 hours/+12 hours)
  Hemorrhage in other areas besides the brain such as the arterial access site or retroperitoneum.

CONTACTS AND LOCATIONS:
Overall Officials: Raul G Nogueira, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ospel JM, Goyal M. A review of endovascular treatment for medium vessel occlusion stroke. J Neurointerv Surg. 2021 Jul;13(7):623-630. doi: 10.1136/neurintsurg-2021-017321. Epub 2021 Feb 26. PMID 33637570
- [Background] Saver JL, Chapot R, Agid R, Hassan A, Jadhav AP, Liebeskind DS, Lobotesis K, Meila D, Meyer L, Raphaeli G, Gupta R; Distal Thrombectomy Summit Group*dagger. Thrombectomy for Distal, Medium Vessel Occlusions: A Consensus Statement on Present Knowledge and Promising Directions. Stroke. 2020 Sep;51(9):2872-2884. doi: 10.1161/STROKEAHA.120.028956. Epub 2020 Aug 6. No abstract available. PMID 32757757
- [Background] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL. Guidelines for the Early Management of Patients With Acute Ischemic Stroke: 2019 Update to the 2018 Guidelines for the Early Management of Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2019 Dec;50(12):e344-e418. doi: 10.1161/STR.0000000000000211. Epub 2019 Oct 30. PMID 31662037
- [Background] Turc G, Bhogal P, Fischer U, Khatri P, Lobotesis K, Mazighi M, Schellinger PD, Toni D, de Vries J, White P, Fiehler J. European Stroke Organisation (ESO) - European Society for Minimally Invasive Neurological Therapy (ESMINT) Guidelines on Mechanical Thrombectomy in Acute Ischaemic StrokeEndorsed by Stroke Alliance for Europe (SAFE). Eur Stroke J. 2019 Mar;4(1):6-12. doi: 10.1177/2396987319832140. Epub 2019 Feb 26. PMID 31165090
- [Background] Campbell BCV, Ma H, Ringleb PA, Parsons MW, Churilov L, Bendszus M, Levi CR, Hsu C, Kleinig TJ, Fatar M, Leys D, Molina C, Wijeratne T, Curtze S, Dewey HM, Barber PA, Butcher KS, De Silva DA, Bladin CF, Yassi N, Pfaff JAR, Sharma G, Bivard A, Desmond PM, Schwab S, Schellinger PD, Yan B, Mitchell PJ, Serena J, Toni D, Thijs V, Hacke W, Davis SM, Donnan GA; EXTEND, ECASS-4, and EPITHET Investigators. Extending thrombolysis to 4.5-9 h and wake-up stroke using perfusion imaging: a systematic review and meta-analysis of individual patient data. Lancet. 2019 Jul 13;394(10193):139-147. doi: 10.1016/S0140-6736(19)31053-0. Epub 2019 May 22. PMID 31128925
- [Background] Ospel JM, Menon BK, Demchuk AM, Almekhlafi MA, Kashani N, Mayank A, Fainardi E, Rubiera M, Khaw A, Shankar JJ, Dowlatshahi D, Puig J, Sohn SI, Ahn SH, Poppe A, Calleja A, Hill MD, Goyal M. Clinical Course of Acute Ischemic Stroke Due to Medium Vessel Occlusion With and Without Intravenous Alteplase Treatment. Stroke. 2020 Nov;51(11):3232-3240. doi: 10.1161/STROKEAHA.120.030227. Epub 2020 Oct 19. PMID 33070714
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] Menon BK, Hill MD, Davalos A, Roos YBWEM, Campbell BCV, Dippel DWJ, Guillemin F, Saver JL, van der Lugt A, Demchuk AM, Muir K, Brown S, Jovin T, Mitchell P, White P, Bracard S, Goyal M. Efficacy of endovascular thrombectomy in patients with M2 segment middle cerebral artery occlusions: meta-analysis of data from the HERMES Collaboration. J Neurointerv Surg. 2019 Nov;11(11):1065-1069. doi: 10.1136/neurintsurg-2018-014678. Epub 2019 Apr 11. PMID 30975736
- [Background] Haussen DC, Lima A, Nogueira RG. The Trevo XP 3x20 mm retriever ('Baby Trevo') for the treatment of distal intracranial occlusions. J Neurointerv Surg. 2016 Mar;8(3):295-9. doi: 10.1136/neurintsurg-2014-011613. Epub 2015 May 6. PMID 25948592
- [Background] Haussen DC, Al-Bayati AR, Eby B, Ravindran K, Rodrigues GM, Frankel MR, Nogueira RG. Blind exchange with mini-pinning technique for distal occlusion thrombectomy. J Neurointerv Surg. 2020 Apr;12(4):392-395. doi: 10.1136/neurintsurg-2019-015205. Epub 2019 Aug 31. PMID 31473647
- [Background] Perez-Garcia C, Moreu M, Rosati S, Simal P, Egido JA, Gomez-Escalonilla C, Arrazola J. Mechanical Thrombectomy in Medium Vessel Occlusions: Blind Exchange With Mini-Pinning Technique Versus Mini Stent Retriever Alone. Stroke. 2020 Nov;51(11):3224-3231. doi: 10.1161/STROKEAHA.120.030815. Epub 2020 Oct 19. PMID 33070712
- [Background] Grossberg JA, Rebello LC, Haussen DC, Bouslama M, Bowen M, Barreira CM, Belagaje SR, Frankel MR, Nogueira RG. Beyond Large Vessel Occlusion Strokes: Distal Occlusion Thrombectomy. Stroke. 2018 Jul;49(7):1662-1668. doi: 10.1161/STROKEAHA.118.020567. Epub 2018 Jun 18. PMID 29915125
- [Background] Nogueira RG, Mohammaden MH, Haussen DC, Budzik RF, Gupta R, Krajina A, English JD, Malek AR, Sarraj A, Narata AP, Taqi MA, Frankel MR, Miller TR, Grobelny T, Baxter BW, Bartolini BM, Jenkins P, Estrade L, Liebeskind D, Veznedaroglu E; Trevo Registry Investigators. Endovascular therapy in the distal neurovascular territory: results of a large prospective registry. J Neurointerv Surg. 2021 Nov;13(11):979-984. doi: 10.1136/neurintsurg-2020-016851. Epub 2020 Dec 15. PMID 33323503
- [Background] Goyal M, Ospel JM, Menon BK, Hill MD. MeVO: the next frontier? J Neurointerv Surg. 2020 Jun;12(6):545-547. doi: 10.1136/neurintsurg-2020-015807. Epub 2020 Feb 14. No abstract available. PMID 32060151
- [Background] Seners P, Turc G, Maier B, Mas JL, Oppenheim C, Baron JC. Incidence and Predictors of Early Recanalization After Intravenous Thrombolysis: A Systematic Review and Meta-Analysis. Stroke. 2016 Sep;47(9):2409-12. doi: 10.1161/STROKEAHA.116.014181. Epub 2016 Jul 26. PMID 27462117
- [Background] Menon BK, Al-Ajlan FS, Najm M, Puig J, Castellanos M, Dowlatshahi D, Calleja A, Sohn SI, Ahn SH, Poppe A, Mikulik R, Asdaghi N, Field TS, Jin A, Asil T, Boulanger JM, Smith EE, Coutts SB, Barber PA, Bal S, Subramanian S, Mishra S, Trivedi A, Dey S, Eesa M, Sajobi T, Goyal M, Hill MD, Demchuk AM; INTERRSeCT Study Investigators. Association of Clinical, Imaging, and Thrombus Characteristics With Recanalization of Visible Intracranial Occlusion in Patients With Acute Ischemic Stroke. JAMA. 2018 Sep 11;320(10):1017-1026. doi: 10.1001/jama.2018.12498. PMID 30208455
- [Background] Tian H, Parsons MW, Levi CR, Lin L, Aviv RI, Spratt NJ, Butcher KS, Lou M, Kleinig TJ, Bivard A. Influence of occlusion site and baseline ischemic core on outcome in patients with ischemic stroke. Neurology. 2019 Jun 4;92(23):e2626-e2643. doi: 10.1212/WNL.0000000000007553. Epub 2019 May 1. PMID 31043475
- [Background] Lima FO, Furie KL, Silva GS, Lev MH, Camargo EC, Singhal AB, Harris GJ, Halpern EF, Koroshetz WJ, Smith WS, Nogueira RG. Prognosis of untreated strokes due to anterior circulation proximal intracranial arterial occlusions detected by use of computed tomography angiography. JAMA Neurol. 2014 Feb;71(2):151-7. doi: 10.1001/jamaneurol.2013.5007. PMID 24323077
- [Background] Thomalla G, Simonsen CZ, Boutitie F, Andersen G, Berthezene Y, Cheng B, Cheripelli B, Cho TH, Fazekas F, Fiehler J, Ford I, Galinovic I, Gellissen S, Golsari A, Gregori J, Gunther M, Guibernau J, Hausler KG, Hennerici M, Kemmling A, Marstrand J, Modrau B, Neeb L, Perez de la Ossa N, Puig J, Ringleb P, Roy P, Scheel E, Schonewille W, Serena J, Sunaert S, Villringer K, Wouters A, Thijs V, Ebinger M, Endres M, Fiebach JB, Lemmens R, Muir KW, Nighoghossian N, Pedraza S, Gerloff C; WAKE-UP Investigators. MRI-Guided Thrombolysis for Stroke with Unknown Time of Onset. N Engl J Med. 2018 Aug 16;379(7):611-622. doi: 10.1056/NEJMoa1804355. Epub 2018 May 16. PMID 29766770
- [Background] Ma H, Campbell BCV, Parsons MW, Churilov L, Levi CR, Hsu C, Kleinig TJ, Wijeratne T, Curtze S, Dewey HM, Miteff F, Tsai CH, Lee JT, Phan TG, Mahant N, Sun MC, Krause M, Sturm J, Grimley R, Chen CH, Hu CJ, Wong AA, Field D, Sun Y, Barber PA, Sabet A, Jannes J, Jeng JS, Clissold B, Markus R, Lin CH, Lien LM, Bladin CF, Christensen S, Yassi N, Sharma G, Bivard A, Desmond PM, Yan B, Mitchell PJ, Thijs V, Carey L, Meretoja A, Davis SM, Donnan GA; EXTEND Investigators. Thrombolysis Guided by Perfusion Imaging up to 9 Hours after Onset of Stroke. N Engl J Med. 2019 May 9;380(19):1795-1803. doi: 10.1056/NEJMoa1813046. PMID 31067369
- [Background] Thomalla G, Boutitie F, Ma H, Koga M, Ringleb P, Schwamm LH, Wu O, Bendszus M, Bladin CF, Campbell BCV, Cheng B, Churilov L, Ebinger M, Endres M, Fiebach JB, Fukuda-Doi M, Inoue M, Kleinig TJ, Latour LL, Lemmens R, Levi CR, Leys D, Miwa K, Molina CA, Muir KW, Nighoghossian N, Parsons MW, Pedraza S, Schellinger PD, Schwab S, Simonsen CZ, Song SS, Thijs V, Toni D, Hsu CY, Wahlgren N, Yamamoto H, Yassi N, Yoshimura S, Warach S, Hacke W, Toyoda K, Donnan GA, Davis SM, Gerloff C; Evaluation of unknown Onset Stroke thrombolysis trials (EOS) investigators. Intravenous alteplase for stroke with unknown time of onset guided by advanced imaging: systematic review and meta-analysis of individual patient data. Lancet. 2020 Nov 14;396(10262):1574-1584. doi: 10.1016/S0140-6736(20)32163-2. Epub 2020 Nov 8. PMID 33176180